CLINICAL TRIAL: NCT06981884
Title: The Effect of Motor Imagery Training on Functional Status, Body Awareness, Quality of Life, and Anxiety Levels in Mothers of Children With Physical Disabilities
Brief Title: Motor Imagery as a Supportive Strategy for Caregiving Mothers: A Randomized Controlled Study on Physical and Somatic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Aydan Selen AYDIN, lecturer, Batman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BATMANU-FTR-ASA-01
Record Dates: First submitted 2025-05-07; First posted 2025-05-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Instability
Keywords: Mothers; Disabled child; Motor imagery; Core stabilization; lumbar instability

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind study consisting of 2 groups: experimental and control. The control group received only core stabilization exercises, the experimental group received motor imagery training + core stabilization exercises.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stabilization exercises group (Active Comparator): Group 1: Core stabilization exercise group Participants will be given core stabilization exercises 2 days a week, 45 minutes per session, for 2 months. At the end of 2 months, the outcome measurements will be taken by an evaluator physiotherapist who is not present during the treatment.
  Interventions: Other: core stabilization exercises
- motor imagery training group (Experimental): Group 2: Core stabilization exercise + motor imagery training group Participants will be given core stabilization exercises and motor imagery training 2 days a week, 60 minutes per session, for 2 months. At the end of 2 months, the outcome measurements will be taken by the same evaluator physiotherapist who is not present during the treatment.
  Interventions: Other: core stabilization exercises; Other: motor imagery training group

INTERVENTIONS:
Other: core stabilization exercises — Participants will be given core stabilization exercises 2 days a week, 45 minutes per session, for 2 months. At the end of 2 months, the outcome measurements will be taken by an evaluator physiotherapist who is not present during the treatment.
Other: motor imagery training group — core stabilization exercise + motor imagery training group Participants will be given core stabilization exercises and motor imagery training 2 days a week, 60 minutes per session, for 2 months. Motor imagery training will be applied for 15 minutes immediately after the core stabilization exercisesAt the end of 2 months, the outcome measurements will be taken by the same evaluator physiotherapist who is not present during the treatment
  Arms: motor imagery training group

SUMMARY:
The aim of this study is to examine the effectiveness of core stabilization exercises applied with motor imagery training on motor imagery skills, functional status, body awareness, dynamic balance, quality of life and anxiety level parameters in mothers with physically disabled children within a biopsychosocial framework and to determine whether motor imagery training given in addition to core stabilization training has an effect on these parameters.

DETAILED DESCRIPTION:
Mothers with special needs children provide physical support to their children in every period of their lives, while meeting their daily care and needs, especially in transfer activities. Staying in the same position for a long time, lifting heavy objects disrupts body mechanics, causes negativities in endurance, flexibility, strength and muscle structure, and reduces the quality of life by increasing anxiety and worry levels. Various applications are needed to cope with these problems and support mothers in this sense. It is known that regular exercise has a positive effect on muscle strength, the body's physiological system, general health and reducing pain. In addition, it has been observed as a result of different studies that it has positive effects on reducing fatigue and increasing the ability to cope with depression and high anxiety levels. In recent years, in addition to classical physiotherapy applications in the mentioned parameters, applications in which cognitive participation is important have begun to be used in physiotherapy. The motor imagery approach is a method created to improve function and increase body awareness and quality of life.The aim of this study is to examine the effectiveness of motor imagery training on motor imagery skills, functional status, body awareness, dynamic balance, quality of life and anxiety level parameters in mothers of physically disabled children.

ELIGIBILITY:
Inclusion Criteria:

* The primary caregiver of the disabled child is the mother
* The prone lumbar instability test is (+)
* Not receiving any medical treatment for pain
* Not having any obstacles to exercise
* VAS ≥4 low back pain at baseline

Exclusion Criteria:

* Pregnancy
* History of previous back surgery in the last year
* Having peripheral vascular diseases,radiculopathy, spondylolisthesis, tumor, systemic inflammatory diseases.
* Having cognitive disorders.
* Having central or peripheral neurological disease affecting mobility.
* Having received physical therapy due to back pain in the last 6 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women aged 18-65 (Mothers of physically disabled children)
Enrollment: 40 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 8 weeks
  The Oswestry Disability Index is a valid functional measure for assessing axial LBP. The Turkish validity and reliability study of the questionnaire was conducted by Yakut and colleagues in 2004 (Yakut et al., 2004). The questionnaire reveals the level of functional disability related to activities of daily living (ADL) such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual life and travel. Each disability in ADL is scored between 0 and 5, with 0 indicating no pain and 5 indicating the worst pain imaginable. The scores are then added up and converted to a percentage of the maximum score of 50. The resulting percentage is used to measure the level of disability. The evaluation is made by taking into account the questions answered as follows. Scoring = (Patient's score / Possible maximum score) X 100
Visual Analog Scale | 8 weeks
  The Visual Analog Scale, a subjective assessment of pain intensity, consists of a 100 mm long line. Participants were asked to rate their back pain during activity using basic descriptions from 0 to 10, such as "no pain" and "worst imaginable pain." The participant placed a mark reflecting the pain intensity, and the distance from the left endpoint to the mark was measured in mm.
Algometer | 8 weeks
  Pressure pain thresholds (PPTs) are usually used to measure deep muscular tissue sensitivity in experimental and clinical studies. The PPT is defined as the amount of pressure over a given area in which a steadily increasing non-painful pressure stimulus turns into a painful pressure sensation. The "gold standard" for measuring pressure pain sensitivity is the electronic pressure algometer, which quantifies the application of mechanical pressure.The pressure was increased steadily at a rate of approximately 1 kg/s. The patient was informed to stop when pressure sensitivity turned into pain. Each assessment was repeated 3 times with 10 seconds between measurements, and the mean value of the measurements was recorded as the pressure pain threshold.The test was stopped as soon as the patient reported pain and the force applied was recorded. BASELINE®, Doloriometer was used for PPT assessment.
McGill's core endurance tests | 8 weeks
  McGill's core endurance tests: McGill's tests were Used to examine participants' core endurance. These tests consisted of four positions: the trunk anterior flexor test, the right and left lateral plank, and trunk posterior extensor test. Participants performed one practice trial that lasted a few seconds to confirm correct positioning and then one test trial was recorded per position where the maximum time (seconds) participants could maintain a static Position was measured. The same investigator visually determined the end of all tests to assure reliability of testing. This investigator used the commands 'start' and 'stop' to initiate and conclude the test while an assistant investigator recorded the times using a stopwatch. The order of the four test positions was randomly assigned.
Modified Star Excursion Balance Test | 8 weeks
  The Modified Star Excursion Balance Test is reliable methods commonly used to clinically assess dynamic balance of the lower extremity.The 8 directions in the Star Excursion Balance Test are arranged as 3 directions in the Modified Star Excursion Balance Test.The tape measures were fixed by sticking them to the floor so that the angle between the anterior and posterolateral and posteromedial directions was 135ᵒ; the angle between the posteromedial-posterolateral directions was 90ᵒ. Then, they were asked to reach 3 times for all directions and the average was taken. The test score was calculated with the formula [Average reach distance (cm) / lower extremity length (cm) x 100]
Pressure Biofeedback | 8 weeks
  A pressure biofeedback device (Chatanooga, Australia, 2005) was used to evaluate the activity of the TrA muscle. The pressure biofeedback device is a tool used in practice in the clinic to measure the pressure produced by the TrA muscle during activation, with an emphasis on segmental stabilization . Before the test, all participants were taught the abdominal wall pulling (abdominal hallowing) maneuver. The pressure biofeedback device was fixed at 70 mmHg. For the measurement of TrA muscle activity, the pressure biofeedback device was placed under the abdomen at the level of the anterior superior iliac spine while the patient was in a supine position. The participant was asked to perform the abdominal hallowing maneuver and continue the contraction for 10 seconds. The change in pressure was recorded, and the highest value from 3 trials was taken.
Modified Schober Test | 8 weeks
  alternatives. Learn more Participants' lumbar flexion flexibility was evaluated with the Modified Schober Test. The researcher physiotherapist placed both thumbs on the participant's posterior superior iliac spine and marked the midpoint of the distance between the two points. Then, 10 cm above and 5 cm below this point were determined and marked. After the researcher physiotherapist told the participant to bend forward as much as possible with their knees straight, he measured and recorded the new distance between the lower and upper limit points. The distance difference between the new measurements is used to indicate the amount of lumbar flexion. A difference of 0-5 cm indicates that lumbar flexion flexibility has decreased, while a difference of 10 cm or more indicates that lumbar flexion flexibility has increased. Values between 5-10 cm are considered normal.
Movement Imagery Questionnaire-3 | 8 weeks
  Participants' motor imagery ability was assessed using the Movement Imagery Questionnaire-3.. The survey consists of 3 sub-dimensions: internal visual imagery, external visual imagery and kinesthetic imagery, and includes 12 tasks. Participants were asked to perform these tasks in the visual and kinesthetic imagery type. Each task was first explained, physically performed, then the participant returned to the starting position and imagery was performed according to the visual/kinesthetic imagery type. The participant rated the ease or difficulty of creating an imagery on a 7-point scale. In this scale, 1 means "very difficult to see/feel" and 7 means "very easy to see/feel". The actions performed included the upper extremity, lower extremity and body. When calculating the score, the scores of all sub-dimensions were added separately and averaged by dividing by 4. A higher score indicates better mental imagery ability.
Body Awareness Questionnaire | 8 weeks
  The Body Awareness Questionnaire is a scale that includes physical, emotional and social elements about a person's sensitivity to normal or abnormal body states and processes and questions their sensitivity to physical reactions.The questionnaire consists of four subscales. These are (1) estimation of body reactions, (2) sleep-wake cycle, (3) estimation of the onset of the disease, and (4) attention to changes and reactions in body processes. Participants were asked to score each of the 18 statements on a scale of 1 to 7 (1=Not true for me at all, 7=Very true for me). The maximum score that can be obtained from the questionnaire is 126, and the minimum score is 18. The higher the score, the better the level of body awareness.

SECONDARY OUTCOMES:
SF-36 | 8 weeks
  Participants' quality of life was assessed using the Short Form-36 (SF-36).The Likert-type scale consisting of 36 questions evaluates quality of life in 8 sub-dimensions: physical functionality (10 questions), social functionality (2 questions), physical role restrictions (4 questions), emotional role restrictions (3 questions), mental and spiritual health (5 questions), energy/vitality (4 questions), pain (2 questions), and general health perception (5 questions). The scale score is calculated separately for each sub-scale. The score to be obtained from each sub-dimension ranges from 0 to 100. The closer the score is to 100, the higher the quality of life.
Trait Anxiety Inventory. | 8 weeks
  Participants' anxiety levels were assessed using the Trait Anxiety Inventory.The Turkish validity and reliability study of the scale developed by Spielberger in 1964 was conducted by Öner and Le Compte in 1983. This inventory has two subscales, each consisting of 20 items, namely the trait anxiety level and the state anxiety level. While the State Anxiety Scale assesses the temporary anxiety level of the person under the circumstances they are currently in, the Trait Anxiety Scale assesses the anxiety levels that individuals generally feel and are not related to a specific cause and are not clearly understood by others. A high score on the 4-point Likert-type scale indicates a high level of anxiety. The Trait Anxiety Scale was used in our study. The reason for this was to determine the general level of anxiety felt by mothers of physically disabled children.
International Physical Activity Questionnaire - Short Form | 8 weeks
  The International Physical Activity Questionnaire Short Form (IPAQ Short Form) was used to determine the physical activity levels of the participants. The Turkish validity and reliability of this questionnaire was conducted by Sağlam et al. (2010). The form, consisting of 7 items, provides data on the time spent by the individual in walking, moderate-intensity and vigorous activities. The form asks how many days in the last week and how long each day heavy physical activity, moderate-intensity physical activity and walking were performed. In addition, the time spent inactive (sitting, lying down, etc.) is determined.
  The physical activity level is determined by the MET-minute score. 1 MET is accepted as 3.5 ml/kg/min. MET values are 8.0 MET for heavy activities, 4.0 MET for moderate-intensity activities and 3.3 MET for walking.
  For example, the walking MET-min/week score of a person who walks 30 minutes, 4 days a week;
  It is calculated as 3.3 X 4 X 30 = 396 MET-min/week.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman Fatih Kılınç Özel Eğitim ve Rehabilitasyon Merkezi, Batman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no reason.

REFERENCES:
- [Background] Imamura M, Alfieri FM, Filippo TR, Battistella LR. Pressure pain thresholds in patients with chronic nonspecific low back pain. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):327-336. doi: 10.3233/BMR-150636. PMID 26406214
- [Background] La Touche R, Grande-Alonso M, Cuenca-Martinez F, Gonzalez-Ferrero L, Suso-Marti L, Paris-Alemany A. Diminished Kinesthetic and Visual Motor Imagery Ability in Adults With Chronic Low Back Pain. PM R. 2019 Mar;11(3):227-235. doi: 10.1016/j.pmrj.2018.05.025. Epub 2019 Jan 15. PMID 29908933
- [Background] Vrana A, Hotz-Boendermaker S, Stampfli P, Hanggi J, Seifritz E, Humphreys BK, Meier ML. Differential Neural Processing during Motor Imagery of Daily Activities in Chronic Low Back Pain Patients. PLoS One. 2015 Nov 16;10(11):e0142391. doi: 10.1371/journal.pone.0142391. eCollection 2015. PMID 26569602
- [Background] Salik Sengul Y, Kaya N, Yalcinkaya G, Kirmizi M, Kalemci O. The effects of the addition of motor imagery to home exercises on pain, disability and psychosocial parameters in patients undergoing lumbar spinal surgery: A randomized controlled trial. Explore (NY). 2021 Jul-Aug;17(4):334-339. doi: 10.1016/j.explore.2020.02.001. Epub 2020 Feb 22. PMID 32147444